CLINICAL TRIAL: NCT03260309
Title: The Influence of Perioperative Optimisation to the Primary Hip Arthroplasty Outcomes
Brief Title: The Influence of Perioperative Optimisation to the Hip Arthroplasty Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Karolinska Institutet (Other); Kaunas University of Technology (Other)
Responsible Party: Principal Investigator, Darius Cincikas, Audrius Andrijauskas PhD , principal investigator, clinical professor, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VilniusU
Record Dates: First submitted 2016-02-29; First posted 2017-08-24 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- semi-closed system group (Experimental): Semi-closed loop infusion system tactic. Programmed iv fluid and blood infusion system ,,Belmont Rapid Infuser" and programmable syringe pump for adrenaline infusion.
  Interventions: Procedure: Semi-closed loop infusion system tactic.
- control group (Experimental): Routine infusion therapy tactic
  Interventions: Procedure: Routine infusion therapy tactic

INTERVENTIONS:
Procedure: Semi-closed loop infusion system tactic. — Semi -closed loop infusion system tactic.Use volume loading test twice (before surgery and 12hrs postoperatively). Computer provides advisory hypotension treatment algorithm. Computer provides advisory anemia treatment algorithm. Programmed iv fluid and blood infusions system ,,Belmont Rapid Infuser" and programmable syringe pump for adrenaline infusion.
  Arms: semi-closed system group
Procedure: Routine infusion therapy tactic — Routine re-hydration bolus before surgery. Routine treatment of hypotension. Routine treatment of anemia.
  Arms: control group

SUMMARY:
Success of the hip arthroplasty depends on the measures that optimize perioperative conditions.It is planned to evaluate semi-closed loop system in the hip arthroplasty surgery.

DETAILED DESCRIPTION:
Success of the total hip arthroplasty depends on the measures that optimize perioperative conditions. They increase the emotional stress of the staff and error probability. It is planned to evaluate semi-closed loop infusion system, its adaption for infusion application's influence to near and far treatment outcomes done by prospective randomized clinical trial. This is done by performing total hip arthroplasty. It's expected to evaluate the semi-closed loop system's influence on the doctor's emotional tension during the decision making.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis of the hip undergoing hip arthroplasty with spinal - epidural anesthesia
* Age >50 and <85 years
* ASA (American Society of Anesthesiology Classification) II physical status
* Start of operation no later than 09:00
* Signed informed consent form

Exclusion Criteria:

* Age <50 and >85 yers
* BMI (Body Mass Index) <20 and >40 kg/m2
* ASA I and ASA>II physical status
* History of a bleeding disorder
* Anemia before surgery Hb<110 g/l
* Intravascular fluid infusion within 24 hours before study
* Diabetes mellitus
* Previous open hip surgery
* Psychiatric illness (intake of other psychiatric medication than selective serotonin reuptake inhibitors)
* Alcohol intake 5 U daily
* Contraindication to spinal - epidural anesthesia
* Surgery not by project surgeon
* Start of operation later than 09:00
* Atrial fibrillation
* Narcotic addiction
* History of DVT (Deep Vein Thrombosis), thromboembolic complications, acute cardiac insufficiency
* Participation in the other study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The efficiency of semi-closed loop infusion system | Before the surgery and 12 hrs postoperatively
  Determine the ratio of doctor's approved and rejected computer suggestions

SECONDARY OUTCOMES:
Perioperative blood loss | Before (baseline) the surgery,during surgery and 24hrs postoperatively
  Non-invasive measurement of Hb (Masimo technology). Laboratory hemoglobin determination, evaluation of the bleeding volume
Coagulation activity | Before (baseline) the surgery and 24hrs postoperatively
  Coagulation activity is investigated thromboelastically
Infused fluid and red blood cell volume | Before the surgery and 24hrs postoperatively
  Repeated rehydration bolus (sol.Ringeri 2,5ml/kg), supportive fluid infusion (sol.NaCl 0,9% 1,5 ml/kg/hrs); evaluation of signs of anemia intolerance if Hb < 110 g/l
Wound healing | Within 6 days postoperatively
  Evaluation of wound tissue condition, measurement of drainage fluid volume
Dosage physical exercise sample | Within 6 days postoperatively
  Timed up and go test
Haemodynamic stability | Before (baseline) the surgery and 12 hrs postoperatively
  Invasive measurement of arterial blood pressure
Complications | Within 6 days postoperatively
  Registration of all complications

CONTACTS AND LOCATIONS:
Overall Officials: Andrijauskas Audrius, PhD, Principal Investigator — Vilnius University

IPD SHARING:
Plan to Share IPD: Undecided